CLINICAL TRIAL: NCT00853892
Title: An Open-Label, Randomized, Two-Period, Crossover Study to Evaluate the Relative Bioavailability of a Controlled-Release Test Tablet Formulation of Oxycodone Hydrochloride (40 mg) Compared to an Equivalent Dose of a Commercially Available Reference Drug Product (OxyContin® 40 mg, Purdue Pharma L.P.) in Normal Human Subjects Under Fasting Conditions
Brief Title: Fasting Study of Controlled-Release Oxycodone Hydrochloride 40 mg Tablets and OxyContin® 40 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Herbert Neuman, MD/Chief Medical Officer, Mallinckrodt
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 0595-05-812
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Healthy
Keywords: Healthy Subjects; Bioequivalence
MeSH Terms: interventions — Tablets; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Controlled-Release Oxycodone Hydrochloride 40 mg tablet
  Interventions: Drug: Controlled-Release Oxycodone Hydrochloride 40 mg tablet
- B (Active Comparator): OxyContin® 40 mg tablet
  Interventions: Drug: OxyContin® 40 mg tablet

INTERVENTIONS:
Drug: Controlled-Release Oxycodone Hydrochloride 40 mg tablet — Controlled-Release Oxycodone Hydrochloride 40 mg, single dose fasting
  Arms: A
Drug: OxyContin® 40 mg tablet — OxyContin® 40 mg tablet, single dose fasting
  Arms: B

SUMMARY:
The objective of this open-label, randomized, two-period, crossover study was to evaluate the oral bioavailability of the Mallinckrodt controlled-release test tablet formulation of oxycodone 40 mg compared to an equivalent oral dose of a commercially available controlled-release tablet of oxycodone (OxyContin® 40 mg, Purdue Pharma L.P.) in a test group of healthy subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-lactating females, 18 years of age or older.
2. Female subjects must be postmenopausal for at least one year, surgically sterile, or practicing adequate non-hormonal contraception for at least 3 months prior to and for the duration of study participation. All female subjects will undergo a pregnancy test at screening and at check-in to the clinical study site for every dosing period. The results of the test must be negative for continued participation.
3. Weight must be within 15% of the ideal weight for height and frame, as adopted by the Metropolitan Life Insurance Co., 1999.
4. Qualifying subjects must be in good health and physical condition as determined by a screening medical history obtained within 30 days prior to study start. Subjects should not present with a history of significant past illness expected to affect the investigation.
5. The normal status of subjects will be confirmed by the following procedures:

   1. Laboratory tests (serum chemistry, hematology, urinalysis). A subject with laboratory values that are not within the clinical laboratory's reference range does not qualify, unless specifically accepted (with comment) by the investigator.
   2. Human immunodeficiency virus (HIV), drugs of abuse, alcohol, and hepatitis B and C testing will be performed at screening. Results of these tests must be negative or non-reactive for subjects to qualify for the study. At each check-in to the study site, a urine drug screen will be performed that must be negative for continued participation.
   3. Electrocardiogram: A 12-lead electrocardiogram (ECG) will be obtained for all subjects at screening. Appropriately trained and experienced medical personnel must interpret this ECG. A subject with an ECG that is not within normal range does not qualify, unless specifically accepted (with comment) by the investigator.
6. Subjects must be able to provide written consent and agree to abide by the study requirements.

Exclusion Criteria:

1. History of chronic alcohol, drug, or narcotic abuse.
2. Chronic use of tranquilizers, sedatives, aspirin, antibiotics, or other medications.
3. History or presence of major organ dysfunction.
4. History of malignancy, stroke, or diabetes; cardiac, renal, liver, pulmonary, or severe gastrointestinal disease; or other serious illness.
5. History of anxiety, tension, severe agitation, psychosis, or mental depression.
6. Family history or diagnosis of epilepsy or other seizure disorder.
7. History of acute abdominal or pelvic conditions.
8. History of conditions which might contraindicate or require caution be used in the administration of oxycodone, including renal impairment, hepatobiliary or pancreatic disease, GI obstruction, cardiac disease, obstructive pulmonary disease, acute or severe bronchial asthma, hypercarbia, elevated intracranial pressure, depleted blood volume, paralytic ileus, or allergy to oxycodone, or history of hypersensitivity to any opiate agonist
9. Administration of any other investigational drug during the 30 days prior to enrollment into the study.
10. Subjects who have smoked or used nicotine-containing products within 6 months prior to study entry.
11. Subjects who have donated blood within 30 days prior to study entry, including that withdrawn during the conduct of any other clinical study.
12. Subjects presenting with acute illness.
13. Subjects who have taken prescription drugs within 14 days or over-the-counter medications (including herbal preparations) within 7 days prior to dosing except for standard daily dose multivitamins.
14. Subjects who have a positive Narcan® challenge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-04; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUCf, AUCinf and Cmax | Two-period crossover with blood samples obtained prior to and following each dose at selected times through 36 hours. Washout period between doses was 7 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Bio-Kinetic Clinical Applications, Springfield, Missouri, United States